CLINICAL TRIAL: NCT07216144
Title: Centralized Lung Cancer Screening Engagement in At-Risk Populations (CLEAR)
Brief Title: Centralized Lung Cancer Screening Engagement in At-Risk Populations
Acronym: CLEAR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 25-04028716
Record Dates: First submitted 2025-10-08; First posted 2025-10-14 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer Screening

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outreach arm (Experimental): Individuals in the outreach arm will receive centralized patient outreach for lung cancer screening in addition to usual care.
  Interventions: Behavioral: Centralized patient outreach for lung cancer screening
- Usual care arm (No Intervention): Individuals in the usual care arm will receive usual care and will not receive any outreach contacts (mail or telephone) within 15 months after randomization.

INTERVENTIONS:
Behavioral: Centralized patient outreach for lung cancer screening — Centralized patient outreach for lung cancer screening will be conducted by the lung screening team and will consist of a letter followed by telephone contact. One week following the mail invitation, a senior patient coordinator (SPC) will make telephone contact with individuals to pre-screen eligibility determination based on pack-year smoking history. Up to three telephone contact attempts will be made within two weeks.
  Arms: Outreach arm

SUMMARY:
This study will assess the impact of centralized outreach on lung cancer screening completion among individuals served by Federally Qualified Health Centers.

DETAILED DESCRIPTION:
This will be a two-arm, parallel, pragmatic randomized controlled trial (RCT) to evaluate the effectiveness of a centralized patient outreach strategy in increasing lung cancer screening (LCS) completion among populations served by Federally Qualified Health Centers (FQHCs). This study will randomize individuals potentially eligible for LCS (50-80 years, current or past smokers) to receive centralized patient outreach in addition to usual care (outreach arm) and usual care alone (usual care arm). Individuals assigned to the outreach arm will receive centralized patient outreach from the Lung screening team through a letter followed by up to three attempts of telephone contact. Individuals assigned to the usual care arm will not receive any contact during the study period and the referral for LCS will be made at the treating physician's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50 to 80 years
* Current or past smokers
* Individuals without a recorded LDCT scan within the past year
* Individuals without a prior lung cancer diagnosis
* Active patients of Ryan Health
* Individuals with a mailing address in the New York City area and a phone number on file

Exclusion Criteria:

* Individuals aged less than 50 or above 80 years
* Individuals without smoking history
* Individuals with a recorded LDCT scan within the past year
* Individuals with a prior lung cancer diagnosis
* Individuals without a mailing address in the New York City area or a phone number on file
* Individuals served by one of Ryan Health clinics where the centralized patient outreach was developed

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of individuals completing low-dose CT (LDCT) within 15 months of randomization. | Within 15 months of randomization

SECONDARY OUTCOMES:
LDCT scan findings: Lung Imaging Reporting and Data System (Lung-RADS) | Within 15 months of randomization
  Proportion of individuals with Lung-RADS 1, 2, 3, and 4
LDCT incident findings | Within 15 months of randomization
  Proportion of individuals with incident findings on LDCT (including moderate to severe coronary artery calcification, lung-mediastinal findings, moderate to severe emphysema, and abdominal findings)
Follow-up care | Within 6 months after screening
  Proportion of individuals receiving a biopsy or lung cancer treatment
Average costs of implementing centralized outreach per individual | Within 15 months of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Jialin Mao, MD, PhD, Principal Investigator — Weill Medical College of Cornell University; Bradley B Pua, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data collected during the trial.
Time Frame: 1 year after publication until 6 years after publication
Access Criteria: Researchers who propose a methodologically sound proposal and receive IRB approval